### DETERMINATION OF SERUM FENTANYL LEVELS AFTER USING REFERENCE AND GENERIC TRANSDERMAL FENTANYL PATCHES WITH AND WITHOUT STANDARDIZED HEAT APPLICATION IN HEALTHY HUMAN VOLUNTEERS

**Short title:** The Effect of Heat on Fentanyl Release from Fentanyl Patches in Healthy Adults

# **Clinical Protocol Principal Investigator:**

Wilbur H. Chen, MD, MS

# **U01 Principal Investigator(s):**

Audra L. Stinchcomb (contact), PhD

Hazem E. Hassan, PhD

### **Sponsor:**

Food and Drug Administration

Grant Number: 1U01FD004955-01

Protocol Number: HP-00059884

NCT02486016

Version 8.0

12 June 2017

#### **CLINICAL STUDY STATISTICS**

#### **IVIVC**

For IVIVC, three correlation levels were examined. Level A was selected to use for analysis of the data. Three different (I, II & III) approaches were examined for Level A.

Level A: a point-to point correlation between in vitro and in vivo profiles.

Level B: comparison between in vitro dissolution time and in vivo residence time.

Level C: a single point correlation between in vitro and in vivo parameters (e.g.  $J_{max}$  vs.  $C_{max}$ ).

Approach I: IVPT data, PK-based mathematical equations and in vitro heat effect coefficient  $(H_i)$  were used to predict in vivo concentrations.

• Eq. 1 Prediction while TDS was worn:



• Eq. 2 Prediction after TDS removal:

C.: Predicted in vivo serum concentration

F: Absolute bioavailability for TDS  $F = \frac{AUC_{0-\infty,TDS} \times Dose_{IV}}{AUC_{0-\infty,IV} \times Dose_{TDS}}$ 

R<sub>in</sub>: Rate of input (mean flux during steady-state in IVPT experiments)

H<sub>i</sub>: In vitro heat effect coefficient (composite heat effect during and after heat exposure); ratio of flux values with heat and without heat

CL: Total body clearance obtained from literature/product package information

k: Elimination rate constant obtained from literature/product package information  $(k_1: after IV dose; k_2: after TDS dose)$ 

t: Time after administration of TDS for Eq.1 and time after removal of TDS for Eq. 2

Co: Initial concentration after TDS removal

#### Approach II and III:

- 1. Reconstruct baseline (32°C) profile by combining the non-heat (32°C) portion of each profile from the early and late heat study designs.
- 2. Deconvolute the in vivo baseline concentration vs time profile using Phoenix®.
- 3. Construct an IVIVC model by plotting the fraction permeated in vitro vs the fraction absorbed in vivo.
- 4. Predict the in vivo fraction absorbed using the IVIVC model and IVPT data.

- 5. Convolute the predicted in vivo fraction absorbed data using Phoenix® to obtain concentration vs time profile
- 6. Apply in vitro heat effect coefficient  $H_i$  (Approach II) or the in vivo heat effect coefficient  $H_{ii}$  (Approach III) to the predicted in vivo profile.

Pharmacokinetic parameters of fentanyl used for Approach I, II and III were obtained from:

- Bower et al. Br J Anaesth 1982
- McClain et al. Clin Pharmacol Ther 1980
- Scott et al. J Pharmacol Exp Ther 1986
- Fung et al. J Clin Pharmacol 1980
- Study [NIPTE-U01-MD-2015-001: Transdermal Drug Delivery Systems-Fentanyl] at University of Maryland, Baltimore; *still in progress*
- *F* [absolute bioavailability for TDS] for Duragesic<sup>®</sup> (0.36) and Mylan (0.42) were each determined from study [NIPTE-U01-MD-2015-001: Transdermal Drug Delivery Systems-Fentanyl] at the University of Maryland, Baltimore
- F [absolute bioavailability for TDS] for Apotex was estimated (0.39) by the mean of 0.36 and 0.42, due to lack of available data